CLINICAL TRIAL: NCT00859404
Title: A 12-week Randomized, Double-blind, Parallel Group, Placebo-controlled Dose Range Finding Study to Evaluate the Efficacy of Oglemilast in the Treatment of Stable Mild to Moderate Persistent Asthma
Brief Title: A Clinical Study of Oglemilast in Patients With Mild to Moderate Persistent Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glenmark Pharmaceuticals Europe Ltd. (R&D) (Industry)
Responsible Party: Dr Narendra Maharaj, Glenmark Pharmaceuticals Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GRC 3886-201
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
Keywords: Mild to moderate persistent asthma
MeSH Terms: conditions — Asthma | interventions — oglemilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1. oglemilast (Experimental)
  Interventions: Drug: oglemilast
- 2. oglemilast (Experimental)
  Interventions: Drug: oglemilast
- 3. oglemilast (Experimental)
  Interventions: Drug: oglemilast
- 4. placebo (Placebo Comparator)
  Interventions: Drug: oglemilast

INTERVENTIONS:
Drug: oglemilast — Tablet oglemilast or placebo once a day, for 12 weeks

SUMMARY:
The study is aimed at evaluating efficacy and safety of oglemilast in the treatment of stable mild to moderate persistent asthma. The study involves two weeks of run in period. This is a placebo controlled study. One of the four treatment arms is placebo. The duration of treatment is 12 weeks.

ELIGIBILITY:
Eligibility Criteria:

* Adult patients with a physician-documented diagnosis of chronic, stable, persistent, mild to moderate asthma (clinical symptoms and documented reversibility of airway obstruction, with an FEV1 of 60% to 85% of the predicted value).

The following criteria must be met at the randomisation visit:

* At least 80% compliance during the single-blind placebo run-in period
* FEV1 between 60% and 85% of the predicted value
* Without asthma exacerbation during the run-in period
* Reversibility: patients are required to demonstrate a ≥ 12% increase in FEV1 (with an absolute improvement in FEV1 of at least 200mL) ≥ 10 min and up to 15 minutes after inhalation of 400 μg salbutamol via a spacer
* Any symptom score being ≥ 1 for at least 4 out of the last 7 days of the run-in
* Use of salbutamol for symptom relief on > 2 occasions on at least 4 out of the last 7 days of the run-in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Morning pre-dose FEV1 at day 85 compared with pre-dose FEV1 value at day 1 | 12 weeks

SECONDARY OUTCOMES:
Change from baseline at days 8, 36 and 64 in morning pre-dose FEV1 | Days 8, 36, 64
Change from baseline at days 8, 36 and 64 in morning pre-dose vital capacity (FVC), peak expiratory flow (PEF), forced expiratory flow 25-75% (FEF25-75%) | days 8, 36 and 64
Change from baseline in morning and evening PEF (based on patient diary) | 12 weeks
Change in asthma day time symptom score from baseline at day 85 | 12 weeks
Change in asthma night time symptom score from baseline at day 85 | 12 weeks
Change in number of night time awakenings from baseline at day 85 | 12 weeks
Frequency and the use of rescue (reliever) medication (salbutamol) | 12 weeks
Frequency and severity of asthma exacerbations | 12 weeks
Investigator global impression of change from baseline to day 85 | 12 weeks
Patient global impression of change from baseline to day 85 | 12 weeks
Pharmacokinetic parameters of oglemilast | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Glenmark investigational sites (28), Mumbai, Bangalore Etc, India